CLINICAL TRIAL: NCT02918097
Title: Cost- Effectiveness and Quality of Life Assessment in Bipolar Disorder Depressive Episode
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Federal University of Rio Grande do Sul (Other)
Responsible Party: Principal Investigator, Ana Flávia Barros da Silva Lima, Principal Investigator, Federal University of Rio Grande do Sul
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 09-013/2
Record Dates: First submitted 2016-09-25; First posted 2016-09-28 (Estimated); Results first posted 2020-10-14 (Actual); Last update posted 2020-11-20 (Actual); Status verified 2016-09

CONDITIONS: Bipolar Disorder
Keywords: Cost effectiveness; Bipolar disorder; Depressive episodes; Quality of Life
MeSH Terms: conditions — Bipolar Disorder | interventions — Lithium Carbonate; Sertraline; Nortriptyline; Risperidone

STUDY DESIGN:
Intervention Model Description: This is a pragmatical clinical trial. The patients follow a pre-established algorithm About the participant flow the results the table to indicate the number of participants who received treatment in the whole algoritm, not in each step.
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lithium Carbonate (Experimental): Group Started: Lithium Carbonate (900mg-1500mg)
  Subjects evaluated for responsiveness every 2 weeks. Responsive to treatment patients remain in the same step. Max. step duration of 8 weeks.
  First step: Monotherapy with Lithium (LSL 0.6-0.8). Non responsive patients: 2nd step.
  Second step: Monotherapy with lithium (LSL 1.0-1.2). Non responsive patients: 3rd step.
  Third step: Lithium + Sertraline (50mg-200mg). Non responsive patients: 4th step.
  Fourth step: Lithium + Nortriptyline 100mg. Non responsive patients: 5th step.
  Fifth step: Lithium + Nortriptyline 100mg + Sertraline (100mg-200mg). Non responsive patients: 6th step
  Sixth step: Lithium + Nortriptyline 100mg + Sertraline 200mg + Risperidone (1mg-6mg).
  Interventions: Drug: Lithium Carbonate; Drug: Sertraline; Drug: Nortriptyline; Drug: Risperidone

INTERVENTIONS:
Drug: Lithium Carbonate
  Other Names: Carbolitium
Drug: Sertraline
  Other Names: Zoloft
Drug: Nortriptyline
  Other Names: Pamelor
Drug: Risperidone
  Other Names: Risperdal

SUMMARY:
To evaluate the effectiveness of an algorithm for Bipolar Disorder depressive episodes (BDD) using medications available in the Brazilian Public Healthcare System (SUS). Quality of life assessment of these patients was also employed.

A randomized pragmatic trial was conducted. An algorithm was developed for the treatment of episodes of bipolar disorder depression episodes.

DETAILED DESCRIPTION:
The study design was that of a pragmatic randomized clinical trial to evaluate the effectiveness of treatments for mood disorders in a public healthcare context in the city of Porto Alegre, in southern Brazil. The algorithm was originally developed for the treatment of bipolar disorder depressive episodes by a Delphi panel of experts from psychiatric associations in Brazil. All subjects provided an informed consent form, in writing, in order to participate in the study protocol, which was approved by the institutional ethics committee.

Procedures and measurements of the study:

The subjects under evaluation were selected and they followed the stages defined by the treatment protocol:

1. Sample selection by being referred from the primary healthcare clinics in the municipality;
2. Informative talk about mood disorders and the research, with the informed consent forms being provided to the subjects;
3. Screening for unipolar depression episodes with the use of the Patient Health Questionnaire (PHQ-9), and Hypomanic Symptoms Checklist Brazilian Version (HCL -32-BV);
4. Diagnostic evaluation through the Mini International Neuropsychiatric Interview (MINI) and clinical interview for individuals with positive results in the screening instruments;
5. Baseline and demographic assessments using standardized semi-structured interviews in the first and second visits;
6. In each clinic visit, the severity of the symptoms were evealuated using the Clinical Global Impression Scale (CGI), Hamilton Rating Scale for Depression (HRSD), and Young Manic Rating Scale (YMRS);
7. Biweekly follow-up, changed to monthly after stabilization - with a maximum follow-up period of 52 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. ages between 18 and 65;
2. BD current acute mixed episode;
3. total capacity to understand and respond to self-applied instruments;
4. the presence of symptoms in the last 30 days;
5. abstinence for at least 30 days for drug addicts.

Exclusion Criteria:

1. presence of Organic Brain Syndrome (OBS);
2. pregnancy or lactation;
3. criteria for psychiatric hospitalization. -

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2010-05; Primary Completion 2014-11 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marcelo Fleck, PhD, Principal Investigator — Federal University of Rio Grande do Sul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lima AF, Miguel SR, Cohen M, Zimmermann JJ, Shansis FM, Cruz LN, Ziegelmann PK, Polanczyk CA, Fleck MP. Effectiveness evaluation of mood disorder treatment algorithms in Brazilian public healthcare patients. Braz J Psychiatry. 2018 Jan-Mar;40(1):26-34. doi: 10.1590/1516-4446-2016-2147. Epub 2017 Aug 21. PMID 28832750

RESULTS

PARTICIPANT FLOW:
Groups:
- Lithium Carbonate: Group Started: Lithium Carbonate (900mg-1500mg)
  Subjects evaluated for responsiveness every 2 weeks. Responsive to treatment patients remain in the same step. Max. step duration of 8 weeks.
  First step: Monotherapy with Lithium (LSL 0.6-0.8). Non responsive patients: 2nd step.
  Second step: Monotherapy with lithium (LSL 1.0-1.2). Non responsive patients: 3rd step.
  Third step: Lithium + Sertraline (50mg-200mg). Non responsive patients: 4th step.
  Fourth step: Lithium + Nortriptyline 100mg. Non responsive patients: 5th step.
  Fifth step: Lithium + Nortriptyline 100mg + Sertraline (100mg-200mg). Non responsive patients: 6th step
  Sixth step: Lithium + Nortriptyline 100mg + Sertraline 200mg + Risperidone (1mg-6mg).
  Lithium Carbonate
  Sertraline
  Nortriptyline
  Risperidone
Period: Overall Study
Arm/Group | Lithium Carbonate
Started | 78
Completed | 58 (Primary and secondary outcomes are assessed just at the end of the protocol, not at each step)
Not Completed | 20

BASELINE CHARACTERISTICS:
Arm/Group | Lithium Carbonate
Number analyzed (Participants) | 78
Age, Continuous [Median (Standard Deviation); unit: years] | 40.4 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61
  Male | 17
Region of Enrollment [Number; unit: participants]
  Brazil | 78

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Response to Treatment"
Description: Response to treatment was defined as a 50% reduction from baseline scores in Hamilton Rating Scale for Depression (HRSD)and Young Mania Rating Scale (YMRS) scales HRSD was developed to evaluate and quantify depression.Its abbreviated version,. Scoring is based on the 17-item scale and scores of 0-7 are considered as being normal. The cutoff points are: 8-17 for mild depression,18-24 for moderate depression, and 25 or more for severe depression. The maximum score being 52 on the 17-point scale.
  YMRS is is the most widely used assessment tool for manic symptoms. The scale consists of 11 items .The YMRS follows the style of the Hamilton Rating Scale for Depression (HAM-D) with each item given a severity rating. There are four items that are graded on a 0 to 8 scale (irritability, speech, thought content, and disruptive/agressive behavior), while the remaining seven items are graded on a 0 to 4 scale. Scores of YMRS > 20 generates indicate mania
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Lithium Carbonate
Number analyzed (Participants) | 78
Participants | 65

2. Primary Outcome: Quality of Life Instrument Scores
Description: Quality of Life - WHOQOL -BREF instrument scores
  scores 0-20 . higher scores mean a better outcome.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lithium Carbonate
Number analyzed (Participants) | 78
score on a scale | 10.58 (3.64)

3. Secondary Outcome: Number of Participants With Remission to Treatment
Description: The remission outcome was established as obtaining three consecutive visits with scores of values considered asymptomatic Hamilton Rating Scale for Depression(HRSD <7 points) and Young Mania Rating Scale (YMRS <6 points) during the trial. The subjects that were asymptomatic for at least 6-8 month were considered to be in partial remission and complete if at least 12 months without symptoms, according to Diagnostic and Statistical Manual of Mental Disorders (DSM-IV).
Time Frame: 8 months
Measure: Count of Participants; unit: Participants
Arm/Group | Lithium Carbonate
Number analyzed (Participants) | 78
Participants | 21

ADVERSE EVENTS:
Time Frame: 18 months
Arm/Group | Lithium Carbonate
All-Cause Mortality (participants affected / at risk) | 0/78
Serious Adverse Events (participants affected / at risk) | 0/78
Other Adverse Events (participants affected / at risk) | 0/78

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No